CLINICAL TRIAL: NCT03029780
Title: Phase II, Randomized, Study of Multiple Administration Regimens for Nivolumab Plus Ipilimumab in Subjects With Renal Cell Carcinoma
Brief Title: An Investigational Immuno-Therapy Safety and Efficacy Study of Multiple Administration Regimens for Nivolumab Plus Ipilimumab in Subjects With Renal Cell Carcinoma
Acronym: CheckMate 800
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-800
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Co-Administration (Experimental): Nivolumab and Ipilimumab Co-Administration
  Interventions: Biological: Opdivo; Biological: Yervoy
- Sequential Administration (Experimental): Nivolumab and Ipilimumab Sequential Administration
  Interventions: Biological: Opdivo; Biological: Yervoy

INTERVENTIONS:
Biological: Opdivo — Specified dose on specified days
  Other Names: Nivolumab
Biological: Yervoy — Specified dose on specified days
  Other Names: Ipilimumab

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of different administration regimens of nivolumab plus ipilimumab in subjects with renal cell carcinoma.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Advanced Renal Cell Carcinoma
* Must have full activity or, if limited, must be able to walk and carry out light activities such as light house work or office work
* Must have at least 1 lesion with measurable disease

Exclusion Criteria:

* Subjects with active central nervous system metastases
* Subjects who received prior therapy with checkpoint inhibitor
* Subjects with active, known or suspected autoimmune disease

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2021-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (11):
- United States (4):
  - Cancer Specialists of North FL, Jacksonville, Florida
  - University Of Iowa Hospitals And Clinics, Iowa City, Iowa
  - Levine Cancer Institute, Charlotte, North Carolina
  - Local Institution, Pittsburgh, Pennsylvania
- Australia (5):
  - Local Institution, Waratah, New South Wales
  - Local Institution, Westmead, New South Wales
  - Local Institution, Herston, Queensland
  - Local Institution, Elizabeth Vale, South Australia
  - Local Institution, Malvern, Victoria
- Chile (2):
  - Centro Internacional de Estudios Clinicos, Recoleta, Santiago de Chile
  - Fundacion Arturo Lopez Perez, Santiago, Santiago Metropolitan

REFERENCES:
- [Derived] Menzies AM, Salman P, Frontera OA, Pook D, Hocking CM, Zakharia Y, Gurney H, Gedye C, Goh JC, Telivala B, Grob JJ, Lebbe C, de la Cruz Merino L, Machet L, Neidhardt EM, Qureshi A, Hosein F, Hamuro L, Simsek B, Amin A. Administration of nivolumab plus ipilimumab: Infusion of the fixed-ratio combination versus sequential infusions in two randomized controlled trials of metastatic melanoma (CheckMate 742) and renal cell carcinoma (CheckMate 800). Cancer. 2025 Jul 15;131(14):e35962. doi: 10.1002/cncr.35962. PMID 40614118
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 104 participants were randomized and treated
Groups:
- Arm A: Fixed Ratio Combination: Participants recieve a fixed ratio combination (BMS-986237) of nivolumab and ipilimumab in a 3:1 ratio (nivolumab 3 mg/kg and ipilimumab1 mg/kg) every 3 weeks for 4 doses. Participants will then receive nivolumab 480 mg flat dose infused over 30 minutes every four weeks.
- Arm B: Sequential Combination: Nivolumab 3 mg/kg and ipilimumab 1 mg/kg will be administered sequentially every 3 weeks for up to 4 doses. Participants will then receive nivolumab 480 mg flat dose infused over 30 minutes every four weeks.
Period: Overall Study
Arm/Group | Arm A: Fixed Ratio Combination | Arm B: Sequential Combination
Started | 52 | 52
Completed | 1 | 1
Not Completed | 51 | 51
Not completed — Disease Progression | 20 | 22
Not completed — Study Drug Toxicity | 15 | 11
Not completed — Adverse Event Unrelated to Study Drug | 2 | 3
Not completed — Participant request to discontinue study treatment | 4 | 1
Not completed — Maximum clinical benefit | 1 | 0
Not completed — Participant no longer meets study criteria | 0 | 1
Not completed — Other reasons | 6 | 6
Not completed — Not reported | 1 | 1
Not completed — Death | 2 | 6

BASELINE CHARACTERISTICS:
Population: All treated participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Fixed Ratio Combination | Arm B: Sequential Combination | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: All treated participants
  Years | 62.2 (10.9) | 62.6 (9.9) | 62.4 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All treated participants
  Participants
    Female | 10 | 14 | 24
    Male | 42 | 38 | 80
Race/Ethnicity, Customized [Number; unit: Count of participants] — Population: All treated participants
  Count of participants
    White | 46 | 51 | 97
    Black or African American | 1 | 0 | 1
    Asian | 3 | 0 | 3
    American Indian or Alaska Native | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participant With Adverse Events (AEs) in the Broad Scope MedDRA Anaphylactic Reaction Standardized MedDRA Queries (SMQ) Within 2 Days After Any Dose in the Combination Period
Description: The percentage of participants who experienced at least 1 adverse event in the MedDRA Anaphylactic Reaction broad scope SMQ with onset on the day of or within 2 days after any study therapy infusion during the combination period (Part 1).
Time Frame: From randomization to 2 days following any dose in the combination period (assessed up to November 24th, 2017, approximately 9 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A: Fixed Ratio Combination | Arm B: Sequential Combination
Number analyzed (Participants) | 52 | 52
Percentage of Participants | 11.5 [4.4 to 23.4] | 11.5 [4.4 to 23.4]
Statistical Analysis 1: Comparison: Arm A: Fixed Ratio Combination vs Arm B: Sequential Combination; Test type: Superiority; DIFFERENCE IN INCIDENCE RATES = 0.0, 95% CI 2-sided [-12.3 to 12.3]
Statistical Analysis 2: Comparison: Arm A: Fixed Ratio Combination vs Arm B: Sequential Combination; Test type: Superiority; Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.30 to 3.39]

2. Secondary Outcome: The Percentage of Participant With Adverse Events in the Narrow Scope MedDRA Anaphylactic Reaction Standardized MedDRA Queries (SMQ) Occurring Within 2 Days After Any Dose in the Combination Period
Description: The percentage of participants who experienced at least 1 adverse event in the MedDRA Anaphylactic Reaction narrow scope SMQ with onset on the day of or within 2 days after any study therapy infusion during the combination period (Part 1).
Time Frame: as for outcome 1
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A: Fixed Ratio Combination | Arm B: Sequential Combination
Number analyzed (Participants) | 52 | 52
Percentage of Participants | 0 [0.0 to 6.8] | 0 [0.0 to 6.8]
Statistical Analysis 1: Comparison: Arm A: Fixed Ratio Combination vs Arm B: Sequential Combination; Test type: Superiority; DIFFERENCE IN INCIDENCE RATES = 0.00, 95% CI 2-sided [0.00 to 0.00]

3. Secondary Outcome: The Percentage of Participants With Drug Related Grade 3-5 Adverse Events
Description: The percentage of participants who experienced at least 1 adverse event of Grade 3 or higher, judged to be related to study treatment by the investigator, with onset on or after the first dose of study treatment and within 30 days of the last dose of study treatment. Evaluated using Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 criteria.
Time Frame: From first dose to 30 days after last dose of study therapy (up to approximately 48 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A: Fixed Ratio Combination | Arm B: Sequential Combination
Number analyzed (Participants) | 52 | 52
Percentage of Participants | 48.1 [34.0 to 62.4] | 42.3 [28.7 to 56.8]
Statistical Analysis 1: Comparison: Arm A: Fixed Ratio Combination vs Arm B: Sequential Combination; Test type: Superiority; DIFFERENCE IN INCIDENCE RATES = 5.8, 95% CI 2-sided [-13.3 to 24.8]
Statistical Analysis 2: Comparison: Arm A: Fixed Ratio Combination vs Arm B: Sequential Combination; Test type: Superiority; Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.58 to 2.78]

4. Secondary Outcome: The Percentage of Participants With All Causality Grade 3-5 Adverse Events
Description: The percentage of participants who experienced at least 1 adverse event of Grade 3 or higher with onset on or after the first dose of study treatment and within 30 days of the last dose of study treatment. Evaluated using the NCI CTCAE version 4.0 criteria
Time Frame: From first dose to 30 days after last dose of study therapy (up to approximately 48 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of Particpants
Arm/Group | Arm A: Fixed Ratio Combination | Arm B: Sequential Combination
Number analyzed (Participants) | 52 | 52
Percentage of Particpants | 73.1 [59.0 to 84.4] | 65.4 [50.9 to 78.0]
Statistical Analysis 1: Comparison: Arm A: Fixed Ratio Combination vs Arm B: Sequential Combination; Test type: Superiority; DIFFERENCE IN INCIDENCE RATES = 7.7, 95% CI 2-sided [-10.1 to 25.5]
Statistical Analysis 2: Comparison: Arm A: Fixed Ratio Combination vs Arm B: Sequential Combination; Test type: Superiority; Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.62 to 3.24]

5. Secondary Outcome: Objective Response Rate (ORR)
Description: The percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR). The BOR is defined as the best response designation, as determined by the investigator, recorded between the date of randomization and the date of objectively documented progression per RECIST 1.1 or the date of first subsequent anti-cancer therapy, whichever occurs first. For participants without documented progression or subsequent therapy, all available response designations will contribute to the BOR assessment. Complete Response is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10mm. Partial Response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From randomization to the date of objectively documented progression or the date of first subsequent anti-cancer (up to approximately 52 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of Particpants
Arm/Group | Arm A: Fixed Ratio Combination | Arm B: Sequential Combination
Number analyzed (Participants) | 52 | 52
Percentage of Particpants | 50.0 [35.8 to 64.2] | 32.7 [20.3 to 47.1]

6. Secondary Outcome: Progression Free Survival (PFS)
Description: The time between the date of randomization and the first date of documented progression, or death due to any cause, whichever occurs first (per investigator). Participants who die without progression will be considered to have progressed on the date of their death. Participants who did not progress or die are censored on the date of their last evaluable tumor assessment. Participants with no on study tumor assessments and who did not die will be censored on their date of randomization. Participants who started anti-cancer therapy without a prior reported progression will be censored on the date of their last evaluable tumor assessment prior to the first subsequent anti-cancer therapy. Progression is defined as at least a 20% increase in the sum of diameters of target lesions. The sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression)
Time Frame: From randomization to the first date of documented progression or death due to any cause (up to approximately 52 months)
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Fixed Ratio Combination | Arm B: Sequential Combination
Number analyzed (Participants) | 52 | 52
Months | 12.06 [9.92 to 18.23] | 7.69 [3.42 to 11.33]

7. Secondary Outcome: Geometric Mean Trough Concentrations of Nivolumab and Ipilimumab
Description: Serum concentration-time data of nivolumab and ipilimumab administered as a fixed ratio combination to that of sequentially administered nivolumab and ipilimumab is summarized prior to the next dose (predose). 1 Cycle = 3 weeks
Time Frame: pre-dose on day 1 of cycle 2 and 4
Population: All treated participants with available serum time-concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Arm A: Fixed Ratio Combination | Arm B: Sequential Combination
Number analyzed (Participants) | 50 | 46
ug/mL
  Ipilimumab - Cycle 2 Day 1: number analyzed (Participants) | 50 | 44
  Ipilimumab - Cycle 2 Day 1 | 3.92 (28.9) | 3.43 (43.1)
  Ipilimumab - Cycle 4 Day 1: number analyzed (Participants) | 45 | 41
  Ipilimumab - Cycle 4 Day 1 | 5.90 (37.8) | 5.39 (39.8)
  Nivolumab - Cycle 2 Day 1 | 16.2 (29.1) | 16.1 (46.3)
  Nivolumab - Cycle 4 Day 1: number analyzed (Participants) | 45 | 41
  Nivolumab - Cycle 4 Day 1 | 28.5 (35.3) | 30.5 (43.1)

8. Secondary Outcome: Geometric Mean End of Infusion (EOI) Concentrations of Nivolumab and Ipilimumab
Description: Serum concentration-time data of nivolumab and ipilimumab administered as a fixed ratio combination to that of sequentially administered nivolumab and ipilimumab is summarized at the end of infusion (EOI). 1 Cycle = 3 weeks
Time Frame: EOI on day 1 of cycle 1, 2, and 4
Population: All treated participants with available serum time-concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Arm A: Fixed Ratio Combination | Arm B: Sequential Combination
Number analyzed (Participants) | 52 | 52
ug/mL
  Ipilimumab - Cycle 1 Day 1: number analyzed (Participants) | 49 | 44
  Ipilimumab - Cycle 1 Day 1 | 17.6 (23.7) | 13.4 (61.1)
  Ipilimumab - Cycle 2 Day 1: number analyzed (Participants) | 49 | 44
  Ipilimumab - Cycle 2 Day 1 | 21.4 (24.8) | 15.6 (37.9)
  Ipilimumab - Cycle 4 Day 1: number analyzed (Participants) | 45 | 37
  Ipilimumab - Cycle 4 Day 1 | 24.9 (31.3) | 19.5 (38.5)
  Nivolumab - Cycle 1 Day 1: number analyzed (Participants) | 49 | 51
  Nivolumab - Cycle 1 Day 1 | 57.1 (22.4) | 60.7 (23.0)
  Nivolumab - Cycle 2 Day 1: number analyzed (Participants) | 49 | 46
  Nivolumab - Cycle 2 Day 1 | 70.6 (27.6) | 79.5 (71.9)
  Nivolumab - Cycle 4 Day 1: number analyzed (Participants) | 45 | 39
  Nivolumab - Cycle 4 Day 1 | 85.1 (30.1) | 88.9 (55.1)

ADVERSE EVENTS:
Time Frame: From the date of first dose to 30 days after last dose of study therapy. (up to approximately 48 months) Participants were assessed for All Cause Mortality from their first dose until the study was completed (up to approximately 52 months)
Arm/Group | Arm A: Fixed Ratio Combination | Arm B: Sequential Combination
All-Cause Mortality (participants affected / at risk) | 26/52 | 29/52
Serious Adverse Events (participants affected / at risk) | 27/52 | 25/52
Other Adverse Events (participants affected / at risk) | 49/52 | 48/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Fixed Ratio Combination (N=52) | Arm B: Sequential Combination (N=52)
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Adrenocortical insufficiency acute (Endocrine disorders) | 2 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 1
Hypophysitis (Endocrine disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1
Biliary obstruction (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Achromobacter infection (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Urosepsis (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Embolism (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Fixed Ratio Combination (N=52) | Arm B: Sequential Combination (N=52)
Anaemia (Blood and lymphatic system disorders) | 5 | 3
Eosinophilia (Blood and lymphatic system disorders) | 4 | 3
Leukopenia (Blood and lymphatic system disorders) | 3 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 3
Hyperthyroidism (Endocrine disorders) | 4 | 5
Hypophysitis (Endocrine disorders) | 2 | 4
Hypothyroidism (Endocrine disorders) | 12 | 8
Abdominal pain (Gastrointestinal disorders) | 7 | 3
Constipation (Gastrointestinal disorders) | 3 | 5
Diarrhoea (Gastrointestinal disorders) | 13 | 11
Nausea (Gastrointestinal disorders) | 7 | 4
Vomiting (Gastrointestinal disorders) | 7 | 2
Asthenia (General disorders) | 5 | 5
Fatigue (General disorders) | 24 | 15
Oedema peripheral (General disorders) | 5 | 1
Pyrexia (General disorders) | 2 | 4
Hepatotoxicity (Hepatobiliary disorders) | 5 | 5
Hypersensitivity (Immune system disorders) | 3 | 2
Bronchitis (Infections and infestations) | 1 | 5
Nasopharyngitis (Infections and infestations) | 4 | 3
Upper respiratory tract infection (Infections and infestations) | 8 | 0
Urinary tract infection (Infections and infestations) | 3 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 4 | 0
Alanine aminotransferase increased (Investigations) | 8 | 6
Amylase increased (Investigations) | 11 | 9
Aspartate aminotransferase increased (Investigations) | 7 | 6
Blood alkaline phosphatase increased (Investigations) | 3 | 1
Blood bilirubin increased (Investigations) | 1 | 3
Blood cholesterol increased (Investigations) | 3 | 4
Blood creatinine increased (Investigations) | 10 | 11
Blood glucose increased (Investigations) | 2 | 3
Blood sodium decreased (Investigations) | 1 | 4
Lipase increased (Investigations) | 14 | 11
Weight decreased (Investigations) | 5 | 2
Decreased appetite (Metabolism and nutrition disorders) | 6 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 12 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Headache (Nervous system disorders) | 7 | 6
Syncope (Nervous system disorders) | 3 | 1
Insomnia (Psychiatric disorders) | 3 | 3
Nephropathy toxic (Renal and urinary disorders) | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 15 | 15
Rash (Skin and subcutaneous tissue disorders) | 20 | 10
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 3
Hypotension (Vascular disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication

DOCUMENTS (2):
  • Study Protocol (2017-08-02): https://cdn.clinicaltrials.gov/large-docs/80/NCT03029780/Prot_001.pdf
  • Statistical Analysis Plan (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT03029780/SAP_000.pdf